CLINICAL TRIAL: NCT04598880
Title: Comparison of 1 Liter PEG With Ascorbate and Sodium Picosulfate / Magnesium Citrate for High Quality Colon Cleansing
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/9317
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-10

CONDITIONS: Colonic Diseases
Keywords: Colonoscopy
MeSH Terms: conditions — Colonic Diseases | interventions — Polyethylene Glycols; picosulfate sodium; magnesium citrate

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to 1 of 2 treatment groups with a 1:1 allocation using block sizes of 6 cases in each center.
Who Masked: Outcomes Assessor
Masking Description: The assignment of each treatment will be displayed at the time of patient enrollment and will be open to the participant and the physician. The investigator who performs the colonoscopy and assesses the primary outcome (digestive endoscopist) is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pleinvue (Experimental): Subjects receive polyethylene glycol + ascorbate (PEG1A) as laxative treatment for colonoscopy preparation.
  Interventions: Drug: Polyethylene glycol + ascorbate
- Citrafleet (Experimental): Subjects receive sodium picosulfate + magnesium citrate (PSCM) as laxative treatment for colonoscopy preparation.
  Interventions: Drug: Sodium picosulfate + magnesium citrate

INTERVENTIONS:
Drug: Polyethylene glycol + ascorbate — Pleinvue® is administered orally in 2 doses (3 sachets) as per SmPC within the previous 18 hours to colonoscopy intervention. First dose is administered at 9 pm on the day before intervention (sachet 1: MACROGOL 3350 100 g + SODIUM SULFATE ANHYDROUS 9 g + SODIUM CHLORIDE 2 g + POTASSIUM CHLORIDE 1 g). Second dose is administered 5 hours before intervention and it is composed by 2 sachets (sachet A: MACROGOL 3350 40 g + SODIUM CHLORIDE 3,2 g + POTASSIUM CHLORIDE 1,2 g; sachet B: SODIUM ASCORBATE 48,11 g + ASCORBIC ACID 7,54 g).
  Other Names: Pleinvue®; PEG1A
  Arms: Pleinvue
Drug: Sodium picosulfate + magnesium citrate — Citrafleet® is administered orally in 2 doses (2 sachets) as per SmPC within the previous 18 hours to colonoscopy intervention. First dose (sachet 1) is administered at 9 pm on the day before intervention. Second dose (sachet 2) is administered 5 hours before intervention. Sachets 1 and 2 have the same composition: SODIUM PICOSULFATE 10 mg + MAGNESIUM OXIDE 3,5 g + CITRIC ACID 10,97 g.
  Other Names: Citrafleet®; PSCM
  Arms: Citrafleet

SUMMARY:
Background:

Colorectal cancer is the most frequent neoplasm and the second cause of cancer death in Spain. Colon cleansing is critical for visualization of lesions at colonoscopy. High-quality cleansing allows for correct detection and resection of all lesions and may contribute to adequate risk stratification and follow-up interval.

Low-volume laxatives improve tolerance of the colonoscopy preparation without reducing its effectiveness. Currently, the most widely used low-volume laxatives are one liter of Polyethylene glycol + ascorbate (PEG1A) and sodium picosulfate + magnesium citrate (PSCM).

The evidence on the comparison of laxatives to achieve a high-quality colonic cleansing is very scarce.

Hypothesis:

Polyethylene glycol 1 liter with ascorbate is superior to sodium picosulfate and magnesium citrate in high-quality colon cleansing.

Objective:

Overall objective:

To compare the global high-quality cleansing frequency between the two laxatives using the Harefield Scale (HS).

The primary objective is to demonstrate non-inferiority in global high-quality cleansing of PEG1A compared to PSCM. If non-inferiority is demonstrated, superiority of PEG1A will be analyzed.

Specific objectives:

* Frequency of global high-quality cleansing using the Boston Bowel Preparation Scale (BBPS).
* Frequency of adequate-quality cleansing using the HS and BBPS scales.
* Tolerance and adverse effects of both laxatives.
* Detection of lesions, total adenomas, advanced adenomas, total serrated lesions, advanced serrated lesions and colorectal cancer.
* Detection of neoplastic lesions in the different colon segments (proximal, transverse, descending, sigmoid and rectum).
* Association between detected lesions and the quality of the preparation, according to the HS and BBPS scales.

Methods:

Phase 4, multi-centric, randomized, single-blind (endoscopist), parallel study with two treatment arms: PEG1A (Pleinvue®) and PSCM (Citrafleet®).

DETAILED DESCRIPTION:
This study will be performed in 1104 patients with a scheduled colonoscopy for any indication, who need a bowel preparation for the colonoscopy.

Subjects will be randomly assigned to 1 of 2 treatment groups with a 1:1 allocation using block sizes of 6 cases in each center. The treatment assignment will be open to the participant and the physician. The investigator who performs the colonoscopy and assesses the primary outcome (digestive endoscopist) will be blinded.

In both treatment groups, participants will receive instructions about colonoscopy preparation. Laxative treatment (PEG1A/PSCM) will be administered in two doses, at 9 pm on the day before intervention and 5 hours before colonoscopy, on an outpatient basis.

The day of the colonoscopy appointment will be the final visit of the study. The participant will be asked through a questionnaire about adherence to instructions, tolerance and acceptability to the preparation, and the appearance of side effects. No follow-up period is considered after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with previously scheduled colonoscopy with any indication: screening, follow-up, or symptoms.

Exclusion Criteria:

* Age less than 18 years or more than 85 years
* Hospital admission at the time of colonoscopy
* Partial or total colectomy
* Severe constipation
* Active inflammatory bowel disease
* Severe kidney or liver failure
* Pregnancy or lactation
* Inability to understand the instructions by language barrier or cognitive disorder
* Refusal to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1104 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
High quality of entire colon cleansing according to the HS | At the time of colonoscopy
  High quality cleansing in the entire colon (global) according to the HS, which is defined as all segments with a score of 3 or 4 points.

SECONDARY OUTCOMES:
High quality of segmental colon cleansing according to the HS | At the time of colonoscopy
  High quality cleansing in each segment of colon (segmental) according to the HS, which is defined as a score of 3 or 4 points.
Successful global and segmental colon cleansing according to the HS | At the time of colonoscopy
  Successful cleansing at a global and segmental level according to the HS, which is defined as a segmental score >=2 points, and at a global level, as all segments with a score of >=2 points.
High quality and adequate quality of global and segmental colon cleansing according to the BBPS | At the time of colonoscopy
  High quality cleansing at a segmental level according to the BBPS, which is defined as a score of 3 points, and at a global level, defined as all segments with a score of 3 points.
  Adequate cleansing at segmental level according to the BBPS, which is defined as a segment with a score >=2 points, and at global level, defined as all segments with a score of >=2 points.
Demographic variables | At the screening visit
  Collected through an anamnesis in a structured interview at the beginning of the study.
Variables associated with inadequate colon cleansing | At the screening visit
  Collected through an anamnesis in a structured interview at the beginning of the study.
Variables associated with neoplastic lesions | At the screening visit
  Collected through an anamnesis in a structured interview at the beginning of the study.
Adherence to colonoscopy preparation instructions | Before the colonoscopy
  Collected according to a validated questionnaire before the colonoscopy.
Tolerance and acceptability of the colonoscopy preparation | Before the colonoscopy
  Collected according to a validated questionnaire before the colonoscopy.
Variables on the lesions detected in the colonoscopy | At the time of colonoscopy
  Collected through the colonoscopy report and the anatomopathological analysis of the lesions.
Safety variables | Before the colonoscopy
  The adverse effects of the laxatives administered will be collected before the colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Antonio Alvarez González, MD, PhD, Principal Investigator — Hospital del Mar (Barcelona, Spain); Eduardo Albéniz, MD, PhD, Principal Investigator — Complejo Hospitalario de Navarra (Pamplona, Spain)
Locations (14):
- Spain (14):
  - Hospital de Viladecans, Viladecans, Barcelona
  - Organización Sanitaria Integrada Araba, Alava
  - Hospital de Poniente, Almería
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Virgen de las Nieves, Granada
  - Clínica Universidad de Navarra, Madrid
  - Hospital de la Princesa, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital La Paz, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Costa del Sol, Marbella
  - Hospital Quirón, Málaga
  - Hospital Santa Bárbara, Soria

IPD SHARING:
Plan to Share IPD: No